CLINICAL TRIAL: NCT02854553
Title: Transversus Abdominis Plane Block Alone Versus Transversus Abdominis Plane Block With Rectus Sheath Block as a Postoperative Analgesia in Anterior Abdominal Wall Liposuction Surgery
Brief Title: TAP Block Alone Versus TAPblock With Rectus Sheath Block in Liposuction Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hassan Mohamed Ali, lecturer in anesthesia department Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAP in liposuction
Record Dates: First submitted 2016-07-30; First posted 2016-08-03 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- TAP (Experimental): Transversus abdominis plane block
  Interventions: Procedure: Transversus abdominis plane block
- TAP and rectus sheath block (Experimental): Transversus abdominis plane block with rectus sheath block
  Interventions: Procedure: Transversus abdominis plane block; Procedure: rectus sheath block
- control (No Intervention): no truncal blocks, conventional analgesia

INTERVENTIONS:
Procedure: Transversus abdominis plane block — ultra sound guides Transversus abdominis plane block
  Arms: TAP; TAP and rectus sheath block
Procedure: rectus sheath block — ultrasound guided rectus sheath block
  Arms: TAP and rectus sheath block

SUMMARY:
The transversus abdominis plane (TAP) block is an effective regional nerve block for the anterior abdominal wall. An anesthesiologist typically administers the TAP block preoperatively with ultrasound guidance. It is not yet commonly used during anterior abdominal wall liposuction, where postprocedural pain remains a major concern for patients and surgeons.

DETAILED DESCRIPTION:
The author investigated the feasibility of administering the TAP block under direct vision and compared postoperative narcotic use in patients who received analgesia by TAP block vs with TAP block i addition to rectus sheath block, both performed under direct vision during anterior abdominal wall liposuction.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II, consent,

Exclusion Criteria:

* allergy, coagulopathy, refusal, mentally unstable

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
pain | Three days
  visual analogue scale for pain assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided